CLINICAL TRIAL: NCT00061503
Title: A Double-Masked, Placebo-Controlled, Paired Comparison Study of the Mechanism of Action of TRAVATAN 0.004% in Subjects With Glaucoma or Ocular Hypertension
Brief Title: Mechanism of Action of TRAVATAN 0.004% in Subjects With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-55
Record Dates: First submitted 2003-05-28; First posted 2003-05-30 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost

INTERVENTIONS:
Drug: Travoprost

SUMMARY:
The primary objective of this study is to describe the effect of TRAVATAN 0.004% Ophthalmic Solution on aqueous humor dynamics in subjects with a clinical diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).

ELIGIBILITY:
* Subjects 18 years of age or older
* of either sex
* of any race
* diagnosed with ocular hypertension or open angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Call For Details, Nebraska, United States